CLINICAL TRIAL: NCT04779190
Title: Low-level Laser Therapy Versus Ultrasound Therapy Combined With Exercise in Patients With Subacromial Impingement Syndrome
Brief Title: Physical Therapy in Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ekin Ilke Sen, Assistant Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulU-2017-855
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Low-Level Light Therapy; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-level laser therapy (Experimental): In the low-level laser therapy group, each patient are going to receive low-level laser therapy and cold-pack therapy and perform a home-based exercise program 5 times a week, once a day for 15 sessions.
  Interventions: Device: Low-level laser therapy; Other: Home-based exercise
- Therapeutic ultrasound (Experimental): In the therapeutic ultrasound group, each patient are going to receive therapeutic ultrasound and cold-pack therapy and perform a home-based exercise program 5 times a week, once a day for 15 sessions.
  Interventions: Device: Therapeutic ultrasound; Other: Home-based exercise
- Control (Active Comparator): Participants are going to perform a home-based exercise program and receive cold-pack therapy 5 times a week, once a day for 15 sessions.
  Interventions: Other: Home-based exercise

INTERVENTIONS:
Device: Low-level laser therapy — Gallium-aluminum-arsenide diode laser device
  Arms: Low-level laser therapy
Device: Therapeutic ultrasound — Therapeutic pulsed ultrasound with a frequency of 1 MHz
  Arms: Therapeutic ultrasound
Other: Home-based exercise — Home-based exercises 3 days a week; each exercise comprises one set with 5 repetitions over 4 weeks.

SUMMARY:
The aim of this study is to evaluate the effects of low-level laser therapy (LLLT) and therapeutic ultrasound combined with home-based exercise in comparison with home-based exercise alone in patients with subacromial impingement syndrome (SIS). Participants are going to evaluate before training, and at the 1-month follow-up and 3-month follow-up using the visual analog scale (VAS) scores for pain during activity, at rest, and at night, and the Shoulder Pain and Disability Index (SPADI).

DETAILED DESCRIPTION:
SIS is an important cause of pain and disability and affects activities of daily living. Therefore, a major goal of SIS treatment is to reduce pain and improve upper extremity function. In this prospective, randomized controlled, single-blind, interventional trial, a total of 60 patients with SIS who met the eligibility criteria are going to enrolled in the study. Eligible participants are going to randomly assign to one of the three groups by an independent blinded researcher, using a computer-generated random numbers and allocation ratio of 1:1:1: the LLLT group (LG, n = 20), the ultrasound therapy group (UG, n = 20), and the control group (CG, n = 20). Participants are going to evaluate before training, and at the 1-month follow-up and 3-month follow-up using the visual analog scale (VAS) scores for pain during activity, at rest, and at night, and the Shoulder Pain and Disability Index (SPADI).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of subacromial impingement syndrome based on physical examinations
* Persistent pain in one shoulder for at least 2 months
* No passive shoulder range of motion limitations
* Failure of improvement in pain after analgesic medications

Exclusion Criteria:

* History of malignancy and systemic rheumatic diseases
* Evidence of systemic or local infection
* Presence of major trauma at the affected shoulder
* History of shoulder surgery
* Rotator cuff lesions in the form of either calcific tendinosis or full-thickness tear as confirmed on MRI scanning

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline activity pain score at 1-months and 3-months | Baseline, 1-month, 3-month
  Visual Analogue Scale-Activity pain (0-10 point). Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Change from baseline rest pain score at 1-months and 3-months | Baseline, 1-month, 3-month
  Visual Analogue Scale-Rest pain (0-10 point). Higher scores mean a worse outcome
Change from baseline Shoulder Pain and Disability Index at 1-months and 3-months | Baseline, 1-month, 3-month
  Shoulder Pain and Disability Index (SPADI) measures shoulder pain and shoulder disability. Total score ranges from 0 to 130, where a higher score indicates a worsening status. Each item is scored with the VAS, which ranges from 0 (no pain or no difficulty) to 10 (worst pain imaginable or very difficult, help required)
Change from baseline night pain score at 1-months and 3-months | Baseline, 1-month, 3-month
  Visual Analogue Scale- Night pain (0-10 point). Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nalan Capan, Study Director — Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)